CLINICAL TRIAL: NCT01015378
Title: Natural History of Sigmoid Diverticulitis: The Geneva Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Pascal Gervaz, Department of Surgery, University Hospital and Medical School Geneva SWitzerland
Other Study IDs: CODIGE
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2009-11

CONDITIONS: Diverticulitis
Keywords: Recurrent sigmoid diverticulitis; diverticulitis; Colon; sigmoid; recurrence
MeSH Terms: conditions — Diverticulitis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diverticulitis of the sigmoid colon - first episode
  Interventions: Procedure: laparoscopid sigmoid resection

INTERVENTIONS:
Procedure: laparoscopid sigmoid resection — A second episode of diverticulitis will be treated with IV antibiotics and documented with CT scan and blood tests

SUMMARY:
Aim: This is a longitudinal cohort study to assess long-term clinical outcome of patients who were admitted in our institution for a first episode of uncomplicated sigmoid diverticulitis.

Methods: All patients who were diagnosed with a first episode of sigmoid diverticulitis will be evaluated for inclusion in the study, pending informed consent. Those patients who have evidence of complicated diverticulitis (fistula, abscess) will receive a recommendation to undergo elective sigmoid resection, while those who have a simple attack will be recruited in the cohort. Follow-up will be performed at yearly intervals through telephone interview with the patient. The duration of study is expected to last 10 years (2010-2020), with >50 new patients/year, for a total of >500 patients.

Endpoints:

1. the occurrence of a second episode of diverticulitis
2. severity and outcome of recurrent diverticulitis
3. evolution in digestive symptoms and quality of life (QoL)
4. need for subsequent elective or emergency sigmoid resection

Rationale: This study will help in determining the risk/benefit of the current approach for this common condition, which is to manage patients conservatively with antibiotics and adopt a wait-and-see attitude. Specifically, the following events will be assessed quantitatively:

* the rate of relapse in an urban community.
* the burden of this common disease on QoL and digestive function
* the percentage of patients who may need emergency surgery

DETAILED DESCRIPTION:
Colonic diverticulosis is an increasingly common condition in the Western societies; in our country, a third of the population is affected by the 6th decade and two-thirds by the 9th decade. Fortunately, a majority of patients with diverticulosis remain asymptomatic; diverticulitis, the most common presentation of diverticular disease, has an estimated incidence of 10 patients per 100,000/year.

The diagnosis of sigmoid diverticulitis is usually suspected clinically in a patient presenting with acute lower abdominal pain, associated with an inflammatory syndrome with elevated CRP and/or leukocytes count. The preferred imaging modality to establish definitive diagnosis is computerized tomography (CT) scan with triple (oral, intravenous and intra-rectal) administration of contrast. CT scan may also influence management by demonstrating whether sigmoid diverticulitis is simple (phlegmonous, showing an infiltration of pericolic fat and a thickening of intestinal wall) or complicated (abscess, fistula or peritonitis).

A majority of patients present with simple diverticulitis, and will be conservatively and successfully managed with antibiotics alone. Full colonoscopy is performed eventually, in order to rule out an associated condition, most notably cancer and Crohn's disease. Colonic diverticular disease is usually restricted to the sigmoid colon, and conservative treatment with antibiotics is indicated in cases of a first attack of uncomplicated diverticulitis, the rationale being that a majority of patients treated for a first episode of acute inflammation will eventually recover and have no further problems.

Elective sigmoidectomy is currently recommended in the following clinical situations:

* Patients who had two episodes of uncomplicated diverticulitis.
* Patients who had one episode of complicated (perforated) diverticulitis, with either pericolic of pelvic abscesses (Hinchey stage I and II respectively), fistula formation and/or stenosis.

These guidelines, however, reflect expert consensus rather than scientific evidence; currently, there is no way to predict for each patient the risk for developing subsequent complications and recurrences. Thus, the important question is to determine whether a conservative approach is not simply delaying definitive treatment and expose patients to additional complications and alterations in quality of life.

3. OBJECTIVES

The main objective of this study is to assess the natural history of sigmoid diverticulitis in a cohort of patients living in an urban community, who had radiological and endoscopic evidence of diverticular disease, who benefited initially from adequate antibiotherapy, received dietary counselling, and were followed for a long period of time. In order to do that, we will assess prospectively the following variables:

3.1. Primary endpoints

* Annual rate of recurrent diverticulitis
* Severity and timing of recurrent episodes
* Quality of Life and gastrointestinal symptoms assessed with the GIQLI questionnaire

3.2. Secondary endpoints

* Risk for undergoing emergency surgery
* Surgical morbidity/mortality

ELIGIBILITY:
4.2. Inclusion criteria

* Informed consent
* A first episode of uncomplicated diverticulitis (see definitions), which was documented with CT scan, required hospital admission, and was successfully managed with intravenous antibiotics Or
* A first episode of complicated diverticulitis (Hinchey I or II - see definition), requiring CT scan-guided percutaneous drainage, and successfully managed without surgery in a patient either unfit for, or refusing to undergo elective sigmoid resection Exclusion criteria
* Age < 18 or > 90
* Associated condition of the colon or rectum (cancer, IBD, polyps)
* Patient unable to communicate in French, English or German

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cohort study is designed in order to detect recurrent episodes of diverticulitis in a population of patients who were previously admitted in our institution for a first episode.
  4.1. Study population
  The cohort will consist in the population of patients with CT-scan demonstrated, endoscopy-proven sigmoid diverticulitis who will be admitted in the Department of Surgery of the University Hospital Geneva from January 1st, 2010 to December 31st, 2019. At baseline, participants are between the ages of 18 and 90, and medical information will be updated every year until the end of follow-up, which is December 31st, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-01; Primary Completion 2012-01 (Estimated); Study Completion 2017-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Scarpa CR, Buchs NC, Poncet A, Konrad-Mugnier B, Gervaz P, Morel P, Ris F. Short-term Intravenous Antibiotic Treatment in Uncomplicated Diverticulitis Does Not Increase the Risk of Recurrence Compared to Long-term Treatment. Ann Coloproctol. 2015 Apr;31(2):52-6. doi: 10.3393/ac.2015.31.2.52. Epub 2015 Apr 30. PMID 25960972
- [Derived] Buchs NC, Konrad-Mugnier B, Jannot AS, Poletti PA, Ambrosetti P, Gervaz P. Assessment of recurrence and complications following uncomplicated diverticulitis. Br J Surg. 2013 Jun;100(7):976-9; discussion 979. doi: 10.1002/bjs.9119. Epub 2013 Apr 17. PMID 23592303